CLINICAL TRIAL: NCT04069247
Title: Effectiveness of E-based Cognitive Behavioral Therapy for Insomnia on Improving Mental Health in Chinese Youths With Insomnia: a Large-scale Randomized Control Trial
Brief Title: Effectiveness of eCBT-I on Improving Mental Health in Chinese Youths With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019.044
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Insomnia
Keywords: cognitive behavioral therapy; insomnia; depression; suicide; youth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-based cognitive behavioral therapy for insomnia (e-CBT-I) (Experimental): The e-CBT-I will be delivered by a mobile application (eSleep) developed by BestCare & SuMian BioTech Co., Ltd. which contains a digital, self-paced, and highly interactive programme. It consists of six weekly sessions with animated elements, including an overview of sleep, sleep restriction, stimulus control, cognitive therapy, structured worry time and relapse prevention. Participants will have access to the e-CBT-I treatment for 12 weeks.
  Interventions: Behavioral: e-CBT-I
- E-based health education (e-HE) (Active Comparator): The e-HE, a psychoeducation/information-approach, also consists of six consecutive sessions which contains information about general sleep knowledge, functions of human organs, nutrition, environmental health, brain health, identification and treatments of common diseases, but the contents are not related to any active therapeutic components of cognitive behavioral therapy for insomnia (CBT-I). Participants will have access to the intervention for 12 weeks.
  Interventions: Behavioral: e-HE

INTERVENTIONS:
Behavioral: e-CBT-I — The e-CBT-I will be delivered through a mobile application (eSleep) with a personal password.
  Arms: E-based cognitive behavioral therapy for insomnia (e-CBT-I)
Behavioral: e-HE — The e-HE will be delivered in control though a mobile application (eSleep) with a personal password.
  Arms: E-based health education (e-HE)

SUMMARY:
This study aims to conduct a randomized control trial to validate the treatment effect of e-based cognitive behavioral therapy for Insomnia (e-CBT-I) on insomnia disorder, and explore whether e-CBT-I could prevent depression and suicide in youths with insomnia and subclinical depression. In addition, to further explore the mechanisms underlying the association between insomnia treatments and psychiatric disorders, this study will evaluate whether changes in candidate factors including insomnia symptoms, poor sleep hygiene, sleep-related unhelpful thoughts and maladaptive behaviors, circadian rhythm disruption and chronic sleep deprivation will mediate the effect of e-CBT-I on prevention of depression and suicide.

DETAILED DESCRIPTION:
Previous studies have documented the associations of insomnia with depression and suicide. Currently, researchers have done considerable work to investigate whether e-CBT-I could be effective in improving psychological well-being for adults, and previous studies have confirmed that e-CBT-I is effective in reducing depressive symptoms and suicidal ideation in adult population.

However, such studies have not been established in youths yet. Additionally, it is still unclear that by which mechanisms e-CBT-I might affect mental health, and whether e-CBT-I could reduce the risk of depression and suicide.

This study will be the first specifically designed investigation of the preventive effects of e-CBT-I for depression and suicide in youths, and the first large scale causal test of the relationship between insomnia treatments and psychiatric disorders. The results can be expected to influence care provision for the youth population who are at a life stage of emerging adulthood and vulnerable to psychiatric disorders. Further, because the investigators will be using an e-CBT-I approach, a scalable solution may be demonstrated as both feasible and effective. The findings of this study will show the possibility of developing novel preventive intervention for depression and suicide by targeting insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Native Han youths in Hong Kong and mainland China, aged between15-25
2. A diagnosis of insomnia disorder measured by ICD-10 Classification of Mental and Behavioural Disorders
3. The presence of moderate or severe insomnia measured by a score of 15 or above on ISI
4. The presence of subclinical depression assessed by a score of between 4 and 20 on PHQ-9
5. Access to smartphones
6. Ability to read and understand research protocol

Exclusion Criteria:

1. Shift workers
2. The presence of prominent suicidality (suicide plans and suicide attempts) measured by MINI via telephone interview
3. A reported diagnosis of psychosis, schizophrenia, bipolar disorder, or neurodevelopmental disorders
4. Medical conditions that could cause poor sleep quality and sleep continuity disruption, such as eczema
5. An additional sleep disorder (other than insomnia) that may potentially contribute to a disruption in sleep continuity and quality, such as excessive sleepiness and possible obstructive sleep apnoea
6. The presence of current MDD or a prior episode of MDD within past two months measured by MINI via telephone interview
7. Women during pregnancy or lactation
8. Currently receiving psychological treatment for insomnia provided by a psychologist and/or pharmacological treatment for depression

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 708 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kwok Wing, MBChB, Principal Investigator — Chinese University of Hong Kong; Lin Lu, PhD, Principal Investigator — Peking University Sixth Hospital; Shirley Xin Li, PhD, Study Director — Hong Kong University; Jihui Zhang, PhD, Study Director — Chinese University of Hong Kong; Le Shi, PhD, Study Director — Peking University Sixth Hospital
Locations (2):
- Peking University Sixth Hospital, Beijing, China
- Department of psychiatry, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen SJ, Que JY, Chan NY, Shi L, Li SX, Chan JWY, Huang W, Chen CX, Tsang CC, Ho YL, Morin CM, Zhang JH, Lu L, Wing YK. Effectiveness of app-based cognitive behavioral therapy for insomnia on preventing major depressive disorder in youth with insomnia and subclinical depression: A randomized clinical trial. PLoS Med. 2025 Jan 21;22(1):e1004510. doi: 10.1371/journal.pmed.1004510. eCollection 2025 Jan. PMID 39836656

RESULTS

PARTICIPANT FLOW:
Groups:
- E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I): The e-CBT-I intervention is a digital, self-paced, and interactive insomnia intervention program delivered through smartphone application (esleep: Android: https://sd-oss-cdn.sumian.com/apk/eSleep_1.0.3-release.apk; iOS: Apple App store) that was developed by our research team (Li Chiu Kong Family Sleep Assessment Unit, Department of Psychiatry, The Chinese University of Hong Kong, Hong Kong SAR), and was modified and issued by BestCare & SuMian BioTech Co, Ltd. The Chinese version (simplified Chinese/Mandarin) of the application was designed to adapt for the language background of the participants in China. The program is developed as based on well-established CBT-I treatment protocol and consists of six 20-30 minutes sequential modules unlocked weekly with animated elements, including (1) overview of sleep, (2) sleep restriction, (3) stimulus control, (4) cognitive restructuring (targeting sleep-related dysfunctional cognitions), (5) structured worry time, and (6) relapse prevention (appendix pp 2). Participants had access to the e-CBT-I intervention for 12 weeks, allowing them additional time to complete the intervention in case they were unable to completed it within the initial 6-week period.
- E-based Health Education (e-HE): The control (e-HE) condition was developed by our research team (Li Chiu Kong Family Sleep Assessment Unit, Department of Psychiatry, The Chinese University of Hong Kong, Hong Kong SAR) and issued by BestCare & SuMian BioTech Co, Ltd. according to a psychoeducation/information approach, in order to provide the credibility of the intervention to the participants, and to control for the potential dosing effect of attention and nonspecific components (e.g., expectation and contact hours). The e-HE is a health promotion program with the same contact hours as e-CBT-I which contains information about general sleep knowledge, functions of human organs, nutrition, environmental health, brain health, identification, and treatments of common diseases, while it did not include any active insomnia and depression therapeutic components (appendix pp 2). Each module was unlocked weekly, and participants had access to the program for 12 weeks. The general sleep knowledge session was purposively added in this sleep related RCT to meet the expectation of the participants.
Period: Overall Study
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE)
Started | 354 | 354
Completed | 315 | 319
Not Completed | 39 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE) | Total
Number analyzed (Participants) | 354 | 354 | 708
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (2.0) | 22.2 (1.9) | 22.1 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 205 | 407
  Male | 152 | 149 | 301
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 354 | 354 | 708
Region of Enrollment [Number; unit: participants]
  Hong Kong | 18 | 23 | 41
  China | 336 | 331 | 667
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Insomnia symptoms were measured by Insomnia Severity Index (ISI). ISI is a seven-item self-report measure designed to assess the nature, severity and impact of insomnia, with a higher total score suggesting more severe insomnia symptoms. Scores range from 0 to 28.
  units on a scale | 18.3 (2.7) | 18.3 (2.6) | 18.3 (2.7)
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — Depressive symptoms were measured by Patient Health Questionnaire-9 (PHQ-9). PHQ-9 is a commonly used self-administered questionnaire to assess depressive symptoms and severity, with a higher total score suggesting more severe depressive symptoms. Scores range from 0 to 27.
  units on a scale | 12.1 (3.2) | 12.1 (3.4) | 12.1 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Depressive Disorder
Description: Major depressive disorder will be confirmed by Mini International Neuropsychiatric Interview (MINI).
Time Frame: Up to 12-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE)
Number analyzed (Participants) | 354 | 354
Participants | 37 | 62

2. Secondary Outcome: Change of Depressive Symptoms
Description: Depressive symptoms will be measured by Patient Health Questionnaire-9 (PHQ-9). PHQ-9 is a commonly used self-administered questionnaire to assess depressive symptoms and severity, with a higher total score suggesting more severe depressive symptoms. Scores range from 0 to 27.
Time Frame: Baseline, post-session 2, post-session 4, post-intervention (week 7/at the conclusion of last session), 6- and 12-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE)
Number analyzed (Participants) | 354 | 354
score on a scale
  Baseline | 12.1 (0.2) | 12.1 (0.2)
  Post-session 2 | 7.6 (0.2) | 7.7 (0.2)
  Post-session 4 | 6.1 (0.2) | 7.0 (0.2)
  Post-intervention | 5.1 (0.2) | 6.2 (0.2)
  6-month | 5.4 (0.2) | 6.3 (0.2)
  12-month | 5.5 (0.2) | 6.0 (0.2)

3. Secondary Outcome: Change of Insomnia Symptoms
Description: Insomnia symptoms will be measured by Insomnia Severity Index (ISI). ISI is a seven-item self-report measure designed to assess the nature, severity and impact of insomnia, with a higher total score suggesting more severe insomnia symptoms. Scores range from 0 to 28.
Time Frame: Baseline, post-session 2 (week 3/at the conclusion of session 2), post-session 4 (week 5/at the conclusion of session 4), post-intervention (week 7/at the conclusion of last session), 6- and 12-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE)
Number analyzed (Participants) | 354 | 354
score on a scale
  Baseline | 18.3 (0.2) | 18.3 (0.2)
  Post-session 2 | 11.5 (0.2) | 12.1 (0.2)
  Post-session 4 | 9.0 (0.2) | 10.7 (0.2)
  Post-intervention | 7.3 (0.2) | 9.3 (0.2)
  6-month | 7.2 (0.2) | 8.4 (0.2)
  12-month | 7.3 (0.2) | 8.2 (0.2)

4. Secondary Outcome: Percentage of Participants in Remission of Insomnia Disorder
Description: Insomnia disorder will be confirmed by International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) Classification of Mental and Behavioural Disorders: Diagnostic Criteria for Research.
Time Frame: Post-intervention (week 7/at the conclusion of last session), 6- and 12-month follow-up
Measure: Number; unit: percentage of participants
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE)
Number analyzed (Participants) | 354 | 354
percentage of participants
  Post-intervention | 52 | 28
  6-month | 56 | 44
  12-month | 57 | 48

5. Other Pre Specified Outcome: Change of Anxiety Symptoms
Description: Anxiety symptoms will be measured by Generalised Anxiety Disorder 7-item (GAD-7). GAD-7 is a self-report measure of anxiety severity, with a higher total score suggesting more severe anxiety symptoms. Scores range from 0 to 21.
Time Frame: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE)
Number analyzed (Participants) | 354 | 354
score on a scale
  Baseline | 7.7 (0.2) | 7.9 (0.2)
  Post-session 2 | 5.8 (0.2) | 6.2 (0.2)
  Post-session 4 | 4.6 (0.2) | 5.6 (0.2)
  Post-intervention | 4.0 (0.2) | 4.9 (0.2)
  6-month | 4.3 (0.2) | 5.0 (0.2)
  12-month | 4.4 (0.2) | 4.8 (0.2)

6. Other Pre Specified Outcome: Percentage of Participants With Suicidality
Description: Suicidality which includes suicidal ideation, suicide plans and suicide attempts will be measured by MINI.
Time Frame: Post-intervention (week 7/at the conclusion of last session), 6- and 12-month follow-up
Measure: Number; unit: percentage of participants
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE)
Number analyzed (Participants) | 354 | 354
percentage of participants
  Post-intervention | 15 | 15
  6-month | 19 | 13
  12-month | 14 | 15

7. Other Pre Specified Outcome: Change of Suicidal Ideation
Description: Suicidal ideation will be measured by Beck Scale for Suicide Ideation (BSSI). BSSI is a 19-item self-report measure designed to assess suicidality, with higher total scores representing greater. Scores range from 0 to 38.
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change of Daytime Symptoms
Description: Daytime symptoms will be measured by Multidimensional Fatigue Inventory (MFI). MFI is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change of Sleep-related Thoughts and Behaviors
Description: Sleep-related thoughts and behaviors will be measured by Brief Version of Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16). DBAS-16 is a 16-item self-report measure designed to evaluate a subset of those sleep related cognition, with a higher score indicating more dysfunctional beliefs and attitudes about sleep. The total score is calculated from the average score of all the items on the scale and could range from 0 to 10.
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change of Circadian Rhythms
Description: Circadian rhythms will be measured by reduced version of Horne and Östberg Morningness-Eveningness Questionnaire (rMEQ). The rMEQ is a 5-item self reported measure used to evaluate circadian rhythm and sleep rhythm patterns in individuals. Individuals scored higher than 17 and lower than 12 were classified as morning-type and evening-type, respectively. Individuals scored between 12 and 17 were classified as intermediate-type. Scores range from 4 to 25.
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change of Subjective Sleep Measure (Time in Bed, TIB)
Description: TIB will be estimated by 7-Day Daily Sleep Diary. 7-Day Daily Sleep Diary is a prospective measure that includes the questions to assess bedtime, time to fall asleep, total length of time awake during the night, number of awakenings during the night, final wake time and rise time, time spent in bed, total sleep time, sleep quality during the previous night (rating 0-10).
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change of Subjective Sleep Measure (Total Sleep Time, TST)
Description: TST will be estimated by 7-Day Daily Sleep Diary. 7-Day Daily Sleep Diary is a prospective measure that includes the questions to assess bedtime, time to fall asleep, total length of time awake during the night, number of awakenings during the night, final wake time and rise time, time spent in bed, total sleep time, sleep quality during the previous night (rating 0-10).
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change of Subjective Sleep Measure (Sleep Onset Latency, SOL)
Description: SOL will be estimated by 7-Day Daily Sleep Diary. 7-Day Daily Sleep Diary is a prospective measure that includes the questions to assess bedtime, time to fall asleep, total length of time awake during the night, number of awakenings during the night, final wake time and rise time, time spent in bed, total sleep time, sleep quality during the previous night (rating 0-10).
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change of Subjective Sleep Measure (Wake After Sleep Onset, WASO)
Description: WASO will be estimated by 7-Day Daily Sleep Diary. 7-Day Daily Sleep Diary is a prospective measure that includes the questions to assess bedtime, time to fall asleep, total length of time awake during the night, number of awakenings during the night, final wake time and rise time, time spent in bed, total sleep time, sleep quality during the previous night (rating 0-10).
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change of Subjective Sleep Measure (Sleep Efficiency, SE)
Description: SE will be estimated by 7-Day Daily Sleep Diary. 7-Day Daily Sleep Diary is a prospective measure that includes the questions to assess bedtime, time to fall asleep, total length of time awake during the night, number of awakenings during the night, final wake time and rise time, time spent in bed, total sleep time, sleep quality during the previous night (rating 0-10).
Time Frame: Baseline, post-intervention, 6- and 12-month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Post-intervention (week 7/at the conclusion of last session), 6- and 12-month follow-up.
Arm/Group | E-based Cognitive Behavioral Therapy for Insomnia (e-CBT-I) | E-based Health Education (e-HE)
All-Cause Mortality (participants affected / at risk) | 0/354 | 0/354
Serious Adverse Events (participants affected / at risk) | 0/354 | 0/354
Other Adverse Events (participants affected / at risk) | 0/354 | 0/354

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT04069247/Prot_SAP_000.pdf